CLINICAL TRIAL: NCT00983112
Title: Impact of a Biological Glue (Evicel®) on the Peri Operative Bleeding in Total Knee Prothesis Surgery
Brief Title: Evicel Study on the Peri-operative Bleeding in Total Knee Prothesis Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Mutualiste Chirurgicale de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009-010802-12; 2009-003
Record Dates: First submitted 2009-09-18; First posted 2009-09-23 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Thrombosis
Keywords: Gonarthrosis; Knee prosthesis insertion; Bleeding; Undergoing a total knee prothesis surgery; knee prothesis surgery; Knee arthrosis; Thrombosis
MeSH Terms: conditions — Thrombosis; Osteoarthritis, Knee; Hemorrhage | interventions — Fibrinogen; Thrombin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evicel (Experimental)
  Interventions: Drug: Human Fibrinogen and human thrombin (Evicel)
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium Chlorure (Physiological saline)

INTERVENTIONS:
Drug: Human Fibrinogen and human thrombin (Evicel) — Product to be applied intraoperatively. No further administration will take place after this.
  Other Names: Evicel
  Arms: Evicel
Drug: Sodium Chlorure (Physiological saline) — Sterile concentration, local use.
  Other Names: Physiological saline
  Arms: Placebo

SUMMARY:
Knee prothesis surgery is responsible of a risk of thrombosis and hemorrhage. To prevent thrombosis, patients have systematic anticoagulation after surgery which are responsible of hemorrhage. A local glue which improve local coagulation and have no impact of thrombosis can be a solution to limit hemorrhage. The purpose of this trial is to study the impact of a biological glue administration on the bleeding loss at five days after a total knee prosthesis surgery operation.

DETAILED DESCRIPTION:
The orthopaedic surgeon administers a local pulverisation of the biological glue during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated with or a beneficiary of a social security category:

  * having more than 18 years old
  * having signed the informed consent form
  * having undergone a total knee prosthesis surgery operation

Exclusion Criteria:

* incapacity to understand the protocol
* patient having taken anti-coagulants or clopidogrel 10 days before excepted aspirin to a dose equal or less than 160 mg/day
* women having period so generally women having less than 50 years old
* PT less than 60% and ACT taller than 10 sec
* contra-indications to the drug
* Erytropoietine treatment required before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Study the impact of a biological glue administration on the bleeding loss at Day 5 after a total knee prosthesis surgery operation | Day 5

SECONDARY OUTCOMES:
The rate of cell saver transfusion the surgery day | Day 0
The rate of red blood cell transfusion | Day 1, Day 3, Day 5 and at the hospitalisation end
The hematoma size | Day 1, Day 3, Day 5 and at the hospitalisation end
The site incision state | Day 1, Day 3, Day 5 and at the hospitalisation end
The rest and movement pain | Day 1, Day 3, Day 5 and at the hospitalisation end
The antalgic consumption | Day 1, Day 3, Day 5 and at the hospitalisation end
The functional recovering index | Day 1, Day 3, Day 5, at the hospitalisation end and at 1 month, 3 months and 6 months post-operative
Major rate or clinically significative hemorrhage. | Between Day 1 and the hospitalisation end
Infectious complications. | Between Day 1 and the hospitalisation end
The rate of SUSARs. | Between Day 1 and the end of the study (6 months post-operative)
The rate ot thrombotics events. | Between Day 1 and the hospitalisation end

CONTACTS AND LOCATIONS:
Overall Officials: Denis BAYLOT, Dr, Principal Investigator — Clinique Mutualiste Chirurgicale
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France